CLINICAL TRIAL: NCT04826614
Title: Randomized Clinical Trial Comparing Efficacy of Optimal Treatment and Conventional Treatment for Major Depressive Disorder in Viet Nam
Brief Title: Comparing Efficacy of Optimal Treatment and Conventional Treatment for Major Depressive Disorder in Viet Nam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Nguyen Thuy Phuong, Medical doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNTPhuong
Record Dates: First submitted 2020-01-04; First posted 2021-04-01 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Major Depressive Disorder
Keywords: Viet Nam; HAM-D; optimized treatment
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimized treatment (Experimental): early adjust dose or change drug
  Interventions: Other: optimized treatment
- routine treatment (Active Comparator): slowly adjust dose or change drug
  Interventions: Other: optimized treatment

INTERVENTIONS:
Other: optimized treatment — early adjust dose or change drug

SUMMARY:
Comparison of efficacy treatment (respond, remission) between the optimized treatment group (dose adjustment or early change other drug based on the change of total score HAM-D 17) and the routine treatment group (start with the lowest effective dose and adjust dose slowly) for depressed patients in Viet Nam

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common with a lifetime prevalence about 16 %. MDD is able to be a recurrent and chronic condition. MDD is the second leading cause of disability worldwide. This disorder can reduce an individual's ability to perform at work or school to fulfill family responsibilities and to enjoy almost daily activities. Some evidences suggest that delay in treatment of MDD result in poorer outcome; longer time to remission is associated with residual symptoms, chronic condition, relapse and poorer recovery.

OBJECTIVE:

This study will compare effectiveness of the treatment by using measurement base care, accessing early improvement or lack of improvement to make decisions about regard to dose alteration, switching another antidepressant with standard treatment.

METHOD:

This study is the 8 week randomized controlled trial. Raters blind to protocol and 2 treatment group. This study conduct from March 2021 to March 2022 in UMC hospital, Ho Chi Minh city, Vietnam.

According to DSM criteria 5, 188 outpatient MDD will be recruited, 18-65 year-old, HAM D 17 ≥ 17 score. All patients will have ability to communicate and to provide the written consent. Exclusion criteria are psychotics, OCD, bipolar, suicide attempts in the current major depressive episode, unsuccessful suicide behavior 3 months ago, chronic another medical conditions (diabetes, hypothyroidism, pregnant, epilepsy, kidney failure, stroke, heart failure, liver failure, adrenal insufficiency)

The studied sample is divided into two groups:

Patients receiving standard treatment (group A):

Patients are treated with the minimally effective dose of an antidepressant which can be combined with other classes, for example, low dose antipsychotic medication, mirtazapine, zopiclone, benzodiazepine if insomnia is associated.

Patients are re-examined two times: after 4 weeks and 8 weeks of treatment to re-evaluate clinical symptoms. The current medication can be adjusted or even changed to another drug if it is necessary. This is decided by the assessment of the doctor at that moment.

The HAM-D 17 scale is used to access the patient three times: at the start of treatment, after 4 weeks, and 8 weeks of treatment by an autonomous researcher.

Patients have the right to stop participating in the study at any time and will be admitted to the hospital for treatment if there is a risk of suicide.

Group of patients receiving personalized and optimized treatment (group B):

HAM-D 17 scale is used to assessed patients at the initiation of treatment. Basing on clinical and severity on the HAMD-17 scale, doctors give the medication with the minimally or medium effective dose of an antidepressant corresponding to moderate or severe depression. The treatment can be combined with other groups of drugs such as antipsychotic drugs, mirtazapine, zopiclone, benzodiazepine if insomnia is included.

After 1 week of treatment, patients will be re-assessed with the HAM-D 17 scale. If there is no early improvement (decrease less than 20% of the initial score of HAM-D 17 scales), medication dose will be increased with a condition that the patient tolerates the drug and feel comfortable. Patients who cannot tolerate the current drug will be switched to another drug.

After 2 weeks of treatment, patients will be re-assessed with the HAM-D 17 scale. If there is still no early improvement (decrease less than 20% of the initial score of HAM-D 17 scales), medication dose will be increased again (to maximum dose) with a condition that the patient tolerates the drug and feel comfortable. Patients who cannot tolerate the current drug will be switched to another drug.

After 4 weeks of treatment, patients will be re-assessed with the HAM-D 17 scale. If a patient does not respond to the ongoing treatment (decrease less than 50% of the initial score of HAM-D 17 scales) with the maximum dose of the current antidepressant, he/she will be switch to another antidepressant After 6 weeks of treatment, patients will be re-assessed with the HAM-D 17 scale. If a patient still does not respond to the current treatment (decrease less than 50% of the initial score of HAM-D 17 scales), he/she will be switch to another antidepressant one more time.

After 8 week of treatment, patients will be re-assessed with the HAM-D 17 scale. Patients who do not respond to treatment or do not recover will continue to be treated and monitored in this outpatient clinic.

Patients have the right to stop participating in the study at any time and will be admitted to the hospital for treatment if there is a risk of suicide.

ELIGIBILITY:
Inclusion Criteria:

* New or first recurrent diagnosed as major depression disorder.
* Having total score HAM-D 17 ≥ 17 point

Exclusion Criteria:

* Can not answer the question in HAM-D 17
* Having psychosis, anxiety disorder, obsessive-compulsive disorder
* Having risk of suicide now or 3 months past
* having medical history: diabetes mellitus, hypothyroidism, hypopituitarism, epilepsy, renal failure, heart failure, stroke, myocardial infarction, liver failure, cirrhosis.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Comparison of rate of respond patient between optimization and routine treatment group | 8 weeks
  Rate of responsers has HAMD-17 score decreases over 50 percent in each treatmennt group at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Dung V Do, Study Director — Ho Chi Minh University of Medicine and Pharmacy
Locations (1):
- University Medical Center, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
age, sex